CLINICAL TRIAL: NCT00081757
Title: An Open Protocol For The Compassionate Use of Thalidomide For Patients With Advanced Or Refractory Malignancies
Brief Title: An Open Protocol for the Compassionate Use of Thalidomide
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UARK 98-023
Record Dates: First submitted 2004-04-19; First posted 2004-04-22 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2010-07

CONDITIONS: Multiple Myeloma
Keywords: Advanced; Refractory; Plasmacytoma; Myeloma Proteins
MeSH Terms: conditions — Multiple Myeloma; Plasmacytoma | interventions — Thalidomide

INTERVENTIONS:
Drug: Thalidomide

SUMMARY:
The purpose of this study is to evaluate the use of thalidomide for the treatment of cancer. Patients with many types of cancers will be enrolled because the researchers will also study how the different cancers respond and what kind of side effects patients will experience.

DETAILED DESCRIPTION:
Angiogenesis is a normal, physiological process in the growing embryo, wound healing and ovulation. Progressive recruitments of blood vessels to the tumor site are thought to result in a self perpetuating loop helping to drive the growth of tumors. This new vasculature also allows competent tumor cells to find access to the vascular system and facilitate distant spread of tumor cells. Neovascularization is apparently an absolute prerequisite for physical expansion of solid tumors to grow beyond the volume of about 1-2 mm in diameter. Several molecular and cellular mechanisms have been identified by which tumor parenchyma may exert its angiogenic effect on host endothelial cells. There is also evidence that endothelial cells themselves, like other stromal cells, may act reciprocally to alter the behavior of adjacent tumor cells in a paracrine or cell contact mediated fashion. There is now known to be a diverse family of angiogenic growth factors, foremost among them being basic FGF and VEGF. Several angiogenic peptide genes have been sequenced and cloned. The degree of vascularization has acquired importance as an independent prognostic indicator in various types of solid tumors. More recently, it has been noted that increased angiogenesis may also be an important feature in hematologic malignancies, e.g. leukemia.

ELIGIBILITY:
Inclusion Criteria

* All patients must have a confirmed malignancy which can be classified as locally advanced or distant metastatic disease and must have either 1) failed on standard therapy or 2) have disease for which in the opinion of the investigator, no adequate standard +therapy exists.
* Patients must be 18 years of age or older. Women of childbearing potential must have a negative pregnancy test and fertile women and men must use a medically acceptable means of birth control while on study and for 6 months thereafter.
* Patients must sign an informed consent to participate in this study.
* SWOG Performance status 0-3, unless related to cancer pain.
* Before starting treatment, women of childbearing potential should have a negative pregnancy test performed within 24 hours prior to beginning therapy.
* Pregnancy testing is not required for 1) women who have been post-menopausal for at least 2 years with no menses, 2) women who have had a hysterectomy.
* Patients must have adequate hematologic function as demonstrated by total white blood count > or = 2000/mm3, adequate renal function as demonstrated by serum creatinine < or = 3.0 mg/dl, and adequate hepatic function as demonstrated by bilirubin < or =1.5 mg/dl and transaminases < or =4 x ULN.

Exclusion Criteria

* Patients must not be eligible for any UAMS participating clinical trial of higher priority.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 1998-09; Study Completion 2005-05

PRIMARY OUTCOMES:
The primary objective of this study is to use thalidomide to treat patients with advanced and/or refractory malignancies as part of a defined treatment protocol.

SECONDARY OUTCOMES:
The secondary objective of this study is to collect further basic safety and efficacy data.

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Fassas, MD, Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences/MIRT, Little Rock, Arkansas, United States

REFERENCES:
- See also: Click here for more information about UAMS — http://www.myeloma.uams.edu